CLINICAL TRIAL: NCT06334393
Title: A Phase 1 Double-blind, Randomized, Dose Finding Clinical Trial With an Open-label run-in Part to Assess the Safety and Immunogenicity of an Inactivated, Adjuvanted Whole Zika Virus Vaccine Candidate (VLA1601) in Healthy Flavivirus-naïve Adults Aged 18 to 49 Years
Brief Title: Phase 1 Trial to Assess the Safety and Immunogenicity of an Inactivated, Adjuvanted Whole Zika Virus Vaccine Candidate (VLA1601) in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VLA1601-102
Record Dates: First submitted 2024-03-06; First posted 2024-03-28 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Zika; Zika Virus Infection
Keywords: vaccine; Phase 1
MeSH Terms: conditions — Zika Virus Infection | interventions — 1018 oligonucleotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- VLA1601 Low dose (Experimental)
  Interventions: Biological: VLA1601
- VLA1601 Low dose + CpG 1018® (Experimental)
  Interventions: Biological: VLA1601; Biological: CpG 1018®
- VLA1601 Low dose + 3M-052-AF (Experimental)
  Interventions: Biological: VLA1601; Biological: 3M-052-AF
- VLA1601 Medium dose (Experimental)
  Interventions: Biological: VLA1601
- VLA1601 High dose (Experimental)
  Interventions: Biological: VLA1601

INTERVENTIONS:
Biological: VLA1601 — 0.45mL (milliliter), Day 1 and 29
Biological: CpG 1018® — CpG 1018® will be investigated in combination with VLA1601 Low dose
  Arms: VLA1601 Low dose + CpG 1018®
Biological: 3M-052-AF — 3M-052-AF will be investigated in combination with VLA1601 Low dose
  Arms: VLA1601 Low dose + 3M-052-AF

SUMMARY:
This phase 1 clinical trial consists of an initial open-label sentinel run-in (n=25) and a randomized, double-blind, dose-finding (n=125) investigating three antigen dose levels (low, medium and high) of VLA1601 and bedside mixing of the low-dose formulation with one of the two additional adjuvants (CpG1018®, 3M-052-AF/AP 60-702). VLA1601 will be administered according to a two-dose regimen (i.e., on Day 1 and Day 29).

The primary objective of this trial is to assess the safety and tolerability of the vaccine candidate up to 7 days after each vaccination; and to assess the immune response induced by the vaccine candidate 28 days after the second vaccination. Additionally, safety and immune response of the vaccine candidate will be monitored throughout the trial.

DETAILED DESCRIPTION:
VLA1601 is a second generation, highly purified, inactivated, whole ZIKV vaccine candidate (adsorbed on aluminum hydroxide) designed for active immunization for the prevention of disease caused by the flavivirus ZIKV.

This is a phase 1 trial, consisting of an initial open-label sentinel run-in (n=25) phase and a randomized, double-blind, dose-finding trial (n=125) in flavivirus naïve adults aged 18 to 49 years. In total approximately 150 participants will be vaccinated in this trial.

The trial will investigate three antigen dose levels (low, medium and high) of VLA1601. In addition, CpG 1018® or 3M-052-AF/AP 60-702 are investigated as add-on adjuvants in the low dose group (bedside mixing). Each dose is formulated with alum (aluminum hydroxide) adjuvant.

In each of the five treatment arms 30 participants (each with 5 sentinel/run-in and 25 randomized participants) will be vaccinated. Each participant will receive 2 vaccinations, one on Day 1 and one on Day 29, which will be administered intramuscularly (i.m.) in the deltoid muscle (non-dominant arm). The screening period can last up to 21 days.

The trial began with the vaccination of 25 sentinel participants (5 participants in each of the 5 treatment arms) in a sequential open-label, staggered dose-escalation manner.

Up to approximately 125 participants will be randomized 1:1:1:1:1, stratified by trial site to 5 treatment arms. The injection volume in each treatment arm will be 0.45 mL at each of the 2 vaccinations.

The primary objective of this trial is to assess the safety and tolerability of the vaccine candidate up to 7 days after each vaccination; and to assess the immune response induced by the vaccine candidate 28 days after the second vaccination.

Following a sponsor review of available safety and immunogenicity data up to 6 months after the second vaccination, all sentinels and randomized participants from most favorable treatment arm(s) will be selected for an on-site visit at Day 395 for long-term safety and immunogenicity assessment. All other treatment arms will be followed only by phone-call for the Day 395 assessment of long-term safety.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 49 years of age
* BMI of ≥18.5 and <30 kg/m2
* generally healthy as determined by the investigator's clinical judgement based on medical history, physical examination, and screening laboratory tests.
* If trial participant is of childbearing potential: negative pregnancy test; employ adequate birth control measures up to Day 208.
* Male participant agrees to employ adequate birth control measures up to 90 days after last vaccination.

Key Exclusion Criteria:

Participant

* has a known history of the following flavivirus infection: Zika Virus (ZIKV), Japanese Encephalitis Virus (JEV), Dengue Virus (DENV), Yellow Fever Virus (YFV), West-Nile Virus (WNV), or Tick-Borne Encephalitis Virus (TBEV).
* received or has plans to receive a licensed or investigational flavivirus vaccine during the course of the trial.
* travelled within 4 weeks prior to trial enrollment or has plans to travel to areas (including within the US) with Zika virus (ZIKV), Japanese Encephalitis Virus (JEV), Dengue Virus (DENV) or Yellow Fever Virus (YFV) active transmission/circulation during the course of the trial .
* received active or passive immunization within 4 weeks prior or planned to get such vaccination after any trial-vaccination.
* presents with clinically significant abnormal laboratory values, as determined by the investigator.
* tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* has history of significant cardiovascular, respiratory (including asthma), metabolic, neurological (including Guillain-Barre syndrome [GBS]), psychiatric, hepatic, rheumatic, autoimmune, hematological, gastrointestinal, or renal disorder.
* with known or suspected defect of the immune system that would prevent an immune response to the vaccine.
* received immuno-suppressive therapy within 4 weeks prior to first vaccination. Radiation therapy or immunosuppressive cytotoxic drugs/ monoclonal antibodies in the previous 3 years.
* with a history of severe hypersensitivity reactions or anaphylaxis.
* with a history of any vaccine related contraindicating event .
* with acute febrile infections within two weeks prior to vaccination in this trial.
* donated blood within 4 weeks or received blood-derived products (e.g. plasma) within 12 weeks prior to vaccination in this trial or plans to donate blood or use blood products during the course of the trial.
* has a rash, dermatological condition or tattoos that would, in the opinion of the investigator, interfere with injection site reaction rating.
* presents with clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* is currently enrolled (ICF signed) or has participated in another clinical trial involving an investigational medicinal product (IMP) or device within 4 weeks prior to trial enrollment or is scheduled to participate in another clinical trial involving an IMP or investigational device during the course of this trial.
* has a known or suspected problem with alcohol or drug abuse

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Solicited Adverse Events | 7 days after each vaccination
  frequency of solicited AEs (injection site and systemic reactions)
Solicited Adverse Events | 7 days after each vaccination
  severity of solicited AEs (injection site and systemic reactions)
Neutralizing antibodies against ZIKA virus (ZIKV) | Day 57
  Geometric mean titer (GMT) for neutralizing antibodies against (ZIKV) determined by virus neutralization assay

SECONDARY OUTCOMES:
Solicited Adverse Events | 7 days after any vaccination
  frequency of solicited AEs (injection site and systemic reactions)
Solicited Adverse Events | 7 days after any vaccination
  severity of solicited AEs (injection site and systemic reactions)
Unsolicited AEs | Day 395
  frequency of unsolicited AEs
Unsolicited AEs | Day 395
  severity of unsolicited AEs
Vaccine-related unsolicited AEs | Day 395
  frequency of vaccine-related unsolicited AEs
Vaccine-related unsolicited AEs | Day 395
  severity of vaccine-related unsolicited AEs
Any AEs | Day 395
  severity of any AEs (including solicited and unsolicited AEs)
Any AEs | Day 395
  frequency of any AEs (including solicited and unsolicited AEs)
Any vaccine-related AEs | Day 395
  severity of any vaccine-related AEs (including solicited and unsolicited AEs)
Any Vaccine-related AEs | Day 395
  frequency of vaccine-related AEs (including solicited and unsolicited AEs)
Adverse Events of Special Interest (AESI) | Day 395
  severity of AESI
Adverse Events of Special Interest (AESI) | Day 395
  frequency of AESI
Vaccine-related Adverse Events of Special Interest (AESI) | Day 395
  frequency of vaccine-related AESI
Vaccine-related Adverse Events of Special Interest (AESI) | Day 395
  severity of vaccine-related AESI
Serious Adverse Events (SAE) | Day 395
  frequency of SAEs
Serious Adverse Events (SAE) | Day 395
  severity of SAEs
Vaccine-related Serious Adverse Events (SAE) | Day 395
  frequency of vaccine-related SAEs
Vaccine-related Serious Adverse Events (SAE) | Day 395
  severity of vaccine-related SAEs
ZIKV-specific neutralizing antibodies | up to Day 395 (including Day 1, 15, 29, 43, 208)
  Geometric Mean Titer (GMT) as determined by virus neutralization assay
Seroconversion rate (SCR) | up to Day 395 (including Day 1, 15, 29, 43, 57, 208)
  Rate of participants with seroconversion (SCR defined as proportion of participants achieving a >4-fold increase in neutralizing anti-ZIKV antibody titer from baseline) compared to baseline determined by virus neutralization assay
Geometric Mean Fold Increase (GMFI) | up to Day 395 (including Day 1, 15, 29, 43, 57, 208)
  Geometric Mean Fold Increase compared to baseline determined by virus neutralization assay

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Flourish Research, Chicago, Illinois
  - Velocity Clinical Research, Sioux City, Iowa
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
After trial completion, Valneva may provide access to individual de-identified participant data and related trial documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Trial Report (CTR)) upon request from qualified researchers, and subject to Valneva's review and approval.